CLINICAL TRIAL: NCT03750409
Title: Assessing Feasibility of Prolonged Repetitive Near Infrared Light Stimulation on Cognitive and Behavioral Symptoms in Early to Mid-Stage Dementia
Brief Title: Assessing Feasibility of Prolonged Repetitive Near Infrared Light Stimulation in Early to Mid-Stage Dementia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Quietmind Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 018-209
Record Dates: First submitted 2018-10-16; First posted 2018-11-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mild to Moderate Dementia
Keywords: dementia
MeSH Terms: conditions — Dementia | interventions — Head Protective Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Helmet Active Device (Active Comparator): Patients will be randomized 2:1 ratio to receive either the helmet active device or the helmet sham matched device. EACH device will be delivered with a highly visible tag with either an 'A' or 'B' respective to the study group the patient was randomized to.
  Interventions: Device: Helmet
- Helmet Sham (Sham Comparator): Patients will be randomized 2:1 ratio to receive either the helmet active device or the helmet sham matched device. EACH device will be delivered with a highly visible tag with either an 'A' or 'B' respective to the study group the patient was randomized to.
  Interventions: Device: Helmet

INTERVENTIONS:
Device: Helmet — The portable device covers the head and weighs about 3.5 lb., and is made of light-weight, durable plastic, it is placed on the head with eye panels facing forward. Elastic straps holding the arrays together easily expand to conform to each subjects' head. Patients may notice slight warming of scalp after usage. This warming effect is similar to wearing a regular motorcycle helmet for a similar duration.
  Other Names: Photobiomodulation device

SUMMARY:
This study will gather data to see if infrared and near infrared light frequency can increase the activity of brain cells and provide support for the cell's ability to repair and protect themselves against further damage.

DETAILED DESCRIPTION:
Research suggests that impaired regional cerebral blood flow (rCBF) [flow of blood in certain parts of the brain] plays an important role in dementia. Infrared and near infrared light frequency has been shown to increase the activity of brain cells and provide support for the cell's ability to repair and protect themselves against further damage. This study will evaluate the effects of repeated brief exposure to near infrared light stimulation twice a day on subjects that have problems such as attention span, working memory, strategies of learning and remembering, planning, organizing, self-monitoring, inhibition and flexible thinking for an 8 week period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50-85 years with an independently provided diagnosis of dementia, probable Alzheimer's type.
* Dementia symptoms not greater than early to mid-stage dementia
* Generally healthy as indicated by recent physical examination within the last 6 months
* If labs are available within the last 6 months, renal function, hepatic function, cardiac function should be normal

Exclusion Criteria:

* Diagnosed actively growing intracranial pathology (tumors etc.)
* Misusing illegal substances or alcohol
* Previous history of stroke
* History of aggression or violence
* History of major psychiatric illness
* No underlying CNS pathology (confined to tumor, epilepsy only)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Memory Score | Before first treatment, at 4 weeks and then at 8 weeks.
  Mini Mental State Exam will be performed in beginning of the study (before first treatment), in the middle of the treatment (in 4 weeks) and in the end of treatment (in the end of 8 weeks). This quick assessment will be able to score assessed individuals using 0-30 scoring range. Collected scores will be compared at different time points and any numerical change in score will be evaluated.
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog test) test | Before first treatment, at 4 weeks and then at 8 weeks.
  ADAS-Cog test will be performed in beginning of the study (before first treatment), in the middle of the treatment (in 4 weeks) and in the end of treatment (in the end of 8 weeks) to measure cognition. This comprehensive test will measure patient's ability of language and memory. Test consist of 11 parts and will help to assess baseline and determine cognitive change over period of treatment using patient's ability to answer questions and given score.
Quantitative Electro Encephalography (QEEG) | Before first treatment, at 4 weeks and then at 8 weeks.
  QEEG measurement will be performed in beginning of the study (before first treatment), in the middle of the treatment (in 4 weeks) and in the end of treatment (in the end of 8 weeks). This measurement will use modern analytic software to process activity of the brain during cognitive task in the forms of electrical signals received from the surface of the scalp. Analytical software uses algorithms to assess recorded brain impulses and evaluate brain function, helping to track changes in the brain function due to treatment.
  Waveforms of EEG being assessed:
  1. Delta frequencies (1-4 HZ) are produced during sleep are widespread in the frontal central region. Delta is necessary for sleep and stillness.
  2. Theta frequencies (4-8 HZ) are associated with selective attention, retrieving newly learned information, and preceding sleep. Theta aids creativity and problem solving.
  3. Alpha frequencies (8-12 HZ) appear in the posterior when the eyes are closed. It is associated with idling and

CONTACTS AND LOCATIONS:
Overall Officials: Jason H Huang, MD, Principal Investigator — Baylor Scott and White Healthcare; Marvin H Berman, PhD, Principal Investigator — Quiet Mind Foundation
Locations (2):
- United States (2):
  - Quietmind Foundation, Elkins Park, Pennsylvania
  - Baylor Scott and White Medical Center, Temple, Temple, Texas

IPD SHARING:
Plan to Share IPD: No